CLINICAL TRIAL: NCT06431425
Title: The Electronic Cardiovascular Genetics (eCG) Clinic for Presymptomatic Genetic Counselling: Evaluation of Uptake, Psychological Impact and Satisfaction Among Users
Brief Title: The Electronic Cardiovascular Genetics (eCG) Clinic for Presymptomatic Genetic Counselling
Acronym: eCG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Amsterdam UMC (Other); University Medical Center Groningen (Other); Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Lieke M van den Heuvel, PhD, Principal Investigator, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IMDI104021006
Record Dates: First submitted 2024-05-08; First posted 2024-05-28 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Inherited Cardiac Disease

STUDY DESIGN:
Intervention Model Description: Non-inferiority randomised controlled trial with a parallel group design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital care path (eCG Family Clinic) (Experimental): Individuals included in the intervention group (eCG Family Clinic), will receive an invitation to the DNA-poli platform after the proband adds their email address to the digital clinic at risk relatives list. The eCG Family Clinic serves as the pre-test counseling, afterwards counseling by a healthcare professional can be requested. Subsequently the at-risk relative decides whether to get genetically tested and if the results are communicated via the DNA-poli platform or via telephone.
  Interventions: Behavioral: eCG Family Clinic
- Current clinical practice (No Intervention): Individuals included in the control group, will receive the family letter via the proband. The relative needs to contact their general practitioner to get a referral to the genetic department. The relative sets up an appointment with a genetic counselor. The relative has a face-to-face session with a healthcare professional and will decide during this conversation whether to get genetically tested. When results are in, another face-to-face appointment is set to discuss the result and if applicable, follow-up steps will be discussed.

INTERVENTIONS:
Behavioral: eCG Family Clinic — The DNA-poli is an online tool which is designed as an addition to the current genetic counseling method to make the process more efficient and to increase the uptake without compromising counseling quality. Probands can invite their at-risk family members by entering their email addresses. The family members are invited to the DNA-poli via which they can get all the information needed to make a well-considered decision about genetic testing. The information is provided in different formats, for example via a virtual assistant and via videos, which they can evaluate at their own pace, and which can be reread or rewatched. Afterwards they can request an appointment with a health care professional and make a definite decision about genetic testing.
  Other Names: DNA poli
  Arms: Digital care path (eCG Family Clinic)

SUMMARY:
Inherited cardiovascular conditions generally inherit following an autosomal dominant pattern. When a mutation is detected in the proband, relatives can have predictive DNA testing, and - when they are carrier - be monitored and timely treated if needed. Currently, less than half of relatives attends genetic counselling. With the eCG Family Clinic, an easily accessible virtual clinic which better suits the needs and preferences of relatives will be offered. At the eCG Family Clinic, relatives will receive tailored information to support informed decision-making, a DNA-test at home if desired, and can be referred for local cardiac monitoring if relatives appear to be a carrier. Implementation of the eCG Family Clinic in clinical practice is compared to current practice in this clinical trial.

DETAILED DESCRIPTION:
Background:

Inherited cardiovascular conditions generally inherit following an autosomal dominant pattern. When a mutation is detected in the proband, relatives can have predictive DNA testing, and - when they are carrier - be monitored and timely treated if needed. Currently, less than half of relatives attends genetic counselling. With the eCG Family Clinic, an easily accessible virtual clinic which better suits the needs and preferences of relatives will be offered. At the eCG Family Clinic, relatives will receive tailored information to support informed decision-making, a DNA-test at home if desired, and can be referred for local cardiac monitoring if relatives appear to be a carrier. Implementation of the eCG Family Clinic in clinical practice (intervention group) is compared to current practice (control group) in this clinical trial.

Hypotheses:

It is hypothesized that the eCG Family Clinic can lower practical barriers for at-risk relatives to attend genetic counselling and equally or better suit the needs of probands and relatives in this regard. A higher uptake of presymptomatic counselling in the eCG Family Clinic (intervention) group is expected.

Design:

A non-inferiority randomised controlled trial (RCT) design with two study arms (parallel-group, control- and intervention group) for this study was chosen. In this study, probands, at-risk relatives and genetic healthcare professionals will be recruited for this study. The Medical Ethical Committee of the University Medical Centre Utrecht (UMCU, NedMec) has approved the study design.

Measures:

In this RCT, the following outcome measures will be evaluated: (1) uptake of presymptomatic counselling among at-risk relatives, (2) satisfaction with provided care among healthcare professionals, probands and at-risk relatives, (3) impact on feelings of anxiety and worry among at-risk relatives, (4) time requested for care provision and administration. Uptake of presymptomatic testing will be evaluated using file research. Data on the other outcome measures will be collected using questionnaires. First, probands will be asked to fill out one questionnaire after informing at-risk relatives. In addition, at-risk relatives are asked to fill out a questionnaire twice: (a) shortly after the presymptomatic counselling (time-point 1) and, (b) after two/three months, in which at-risk relatives who chose to have DNA-testing, will have received their results. Finally, healthcare professionals involved in providing counselling will be asked to fill out one questionnaire after study completion. Questionnaires will also be used to administer sociodemographic and clinical characteristics of study participants.

Sample size calculation:

Assuming a two-sided 5% significance level and a power of 80%, 238 at-risk relatives ( 119 per study arm) will be included. Previous literature shows that on average four adult relatives per proband are at 50% risk of inheriting the genetic mutation. Using a conservative estimate of 3.5 relatives per proband, a total of 68 probands (34 per study arm) needs to be included in this study.

Statistical analyses:

Sociodemographic and clinical characteristics will be analysed using descriptive and frequency statistics. Differences in participant characteristics between study arms will assessed with chi-square tests / t-tests, as appropriate. Differences in uptake of genetic counselling will be analysed using chi-square tests; logistic regression analyses will be conducted to assess differences in uptake while controlling for the influence of coviarates. Multilevel analyses will be performed to assess whether the study group has an impact on satisfaction with the care provided and impact on psychological functioning, adjusted for coviarates. SPSS version 29.0.1 will be used to perform statistical analyses. A p-level of p<0.05 will be used.

ELIGIBILITY:
Inclusion Criteria:

Probands:

* > 18 y/o
* Diagnosed with inherited hypertrophic cardiomyopathy (HCM) or dialted cardiomyopathy (DCM))
* Class 4 or 5 variant identified.
* Access to a working laptop or computer device.

At risk relatives:

* > 18 y/o
* First degree family member, or second degree in case of a deceased first degree relative
* Access to a working laptop or computer device.

Healthcare professionals:

- Genetic counsellors of the genetics department directly involved in the care given to the family.

Exclusion Criteria:

- Insufficient control of the Dutch language or digital skills.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Uptake | 1 year post disclosure of the proband result
  Uptake of genetic counselling and predictive DNA testing: i.e., the number of family members attending genetic counselling / pursuing genetic testing, relative to the total number of family members eligible for genetic counselling / genetic testing.
Experience with the eCG Family Clinic | T1: on average 4 weeks, after counselling, T2: on average after 1/2 months, after receiving the DNA test results
  Measured using a self-constructed 9-item questionnaire, with answer options ranging from 1=totally disagree to 5=totally agree (score range: 0-36). In addition, the Dutch patient Satisfaction Questionnaire (PSQ) will be administered among relatives. This questionnaire consists of 5 questions using a 10-point scale (1=not at all to 10=a lot). Scores range from 0-45. A higher score indicates higher satisfaction.

SECONDARY OUTCOMES:
Empowerment / genetic counselling outcomes | T1: on average 4 weeks, after counselling, T2: on average after 1/2 months, after receiving the DNA test results
  Measured using the genetic counseling outcome scale (GCOS). The GCOS consists of 24 questions using a 7-point likert scale (1=totally disagree to 7=totally agree). Total scores range from 0-144, with a higher score indicating higher empowerment.
Informed decision-making | T1: on average 4 weeks, after counselling, T2: on average after 1/2 months, after receiving the DNA test results
  Measured the Decisional Conflict Scale (DSC). The DSC consists of 16 questions using a 5 point Likert Scale (1=totally disagree, to 5= totally agree, total score range 0-64). A higher score indicates higher certainty about the decision made. Furthermore, informed decision-making is measures by 5 self-constructed knowledge questions, which can be answered with 'yes', 'no' or 'I don't know'.
Impact on feelings of anxiety | T1: on average 4 weeks, after counselling, T2: on average after 1/2 months, after receiving the DNA test results
  Measured using the shortened State Trait Anxiety Inventory (STAI). The shortened STAI consists of 6 questions on a 4 point Likert scale (1=not at all, 4=a lot). Total scores range from 0-18, with a higher score indicating higher levels of anxiety.
Efficiency | Administered per genetic consultation through study completion, on average two years
  Measured by administering time needed for counselling / administration per at-risk relative

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Utrecht, Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No